CLINICAL TRIAL: NCT00484536
Title: Double-blind, Placebo-controlled, Randomized, Parallel-group Phase II Study in Subjects With Relapsing Forms of Multiple Sclerosis (MS) to Evaluate the Safety, Tolerability, and Effects of CDP323.
Brief Title: Placebo Controlled Study in Subjects With Relapsing Forms of MS to Evaluate the Safety, Tolerability and Effects of CDP323
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was discontinued due to unfavorable interim analysis
Sponsor: UCB Pharma (Industry)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C32322; 2006-002204-33 (EudraCT Number)
Record Dates: First submitted 2007-06-08; First posted 2007-06-11 (Estimated); Last update posted 2011-09-12 (Estimated); Status verified 2011-03

CONDITIONS: Multiple Sclerosis
Keywords: CDP323; Relapsing Multiple Sclerosis; Magnetic Resonance Imaging; Oral Compound; MS
MeSH Terms: conditions — Multiple Sclerosis | interventions — CDP323

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CDP323 1000 mg/day (Experimental)
  Interventions: Drug: CDP323
- CDP323 500 mg/day (Experimental)
  Interventions: Drug: CDP323
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: CDP323 — 250 mg capsules, 500 mg bid (1000 mg/day)
  Arms: CDP323 1000 mg/day
Drug: placebo — capsules, once daily
  Arms: Placebo
Drug: CDP323 — 250 mg Capsules, 500 mg, once daily
  Arms: CDP323 500 mg/day

SUMMARY:
The objective of the study is to evaluate the effect, safety and tolerability of CDP323 in patients with relapsing forms of multiple sclerosis

ELIGIBILITY:
Inclusion Criteria:

* relapsing form of MS
* screening EDSS score 0 - 5.5, inclusive
* at least one clinical relapse in the 12 months before screening
* active disease, defined by set of MRI activity criteria
* failed prior treatment with beta-interferons or glatiramer acetate

Exclusion Criteria:

* signs of silent infections, including positive tests for HIV1, HIV2 or Hepatitis B or Hepatitis C or tuberculosis
* known allergy to gadolinium-DTPA, and/or ingredients of the study drug formulation
* pre-treatment with immunosuppressive or immunomodulatory drugs prior to screening within certain time frames

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 232 (Actual)
Dates: Start 2007-05; Primary Completion 2009-11 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
The cumulative number of newly active lesions on standardized brain MRI scans after 24 weeks of treatment (Week 28). | Cumulative number of newly active lesions from baseline to Week 28.
  The following lesions are considered newly active: new gadolinium enhancement on T1-weighted images; new lesions on T2-weighted images, but non-enhancing on T1-weighted images; new enlargement on T2-weighted images, but non-enhancing on T1-weighted images.

SECONDARY OUTCOMES:
Occurrence of any treatment emergent adverse event. | During up to 24 weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (71):
- United States (22):
  - Cullman, Alabama
  - Phoenix, Arizona
  - Tucson, Arizona
  - Springs, Colorado
  - Washington D.C., District of Columbia
  - Maitland, Florida
  - Atlanta, Georgia
  - Northbrook, Illinois
  - Fort Wayne, Indiana
  - Kansas City, Kansas
  - Lenexa, Kansas
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Farmington Hills, Michigan
  - Charlotte, North Carolina
  - Columbus, Ohio
  - Providence, Rhode Island
  - Nashville, Tennessee
  - Dallas, Texas
  - Kirkland, Washington
  - Charleston, West Virginia
  - Milwaukee, Wisconsin
- Belgium (6):
  - Diepenbeek
  - Ghent
  - Melsbroek
  - Overpelt
  - Sijsele
  - Sint-Truiden
- Canada (5):
  - London, Ontario
  - Ottawa, Ontario
  - Gatineau, Quebec
  - Greenfield Park, Quebec
  - Sherbrooke, Quebec
- Finland (3):
  - Oulu
  - Tampere
  - Turku
- France (5):
  - Besançon
  - Clermont-Ferrand
  - Lyon
  - Rennes
  - Strasbourg
- Germany (8):
  - Bayreuth
  - Berlin
  - Giessen
  - Hamburg
  - Marburg
  - Rostock
  - Ulm
  - Wiesbaden
- Hungary (4):
  - Budapest
  - Győr
  - Nyíregyháza
  - Pécs
- Netherlands (4):
  - Amsterdam
  - Breda
  - Nieuwegein
  - Nijmegen
- Spain (8):
  - Barcelona
  - Bilbao
  - Girona
  - Madrid
  - Málaga
  - Oviedo
  - Santa Cruz de Tenerife
  - Seville
- Sweden (2):
  - Gothenburg
  - Umeå
- United Kingdom (4):
  - Hartshill
  - Newcastle
  - Nottingham
  - Sheffield